CLINICAL TRIAL: NCT01008696
Title: Effect of Rabeprazole and Lansoprazole on Reflux Esophagitis in Relation to CYP2C19 Genotype Status: A Prospective, Randomized, Multicenter Study
Brief Title: An Efficacy Study to Compare the Treatment Effects of Rabeprazole and Lansoprazole Depending on the Genotyping of CYP2C19 in Treating Reflux Esophagitis
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Janssen Korea, Ltd., Korea (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR013831; RAB-KOR-4023
Record Dates: First submitted 2009-11-05; First posted 2009-11-06 (Estimated); Results first posted 2013-08-13 (Estimated); Last update posted 2013-08-13 (Estimated); Status verified 2013-07

CONDITIONS: Reflux Esophagitis
Keywords: Reflux esophagitis; Rabeprazole; Lansoprazole
MeSH Terms: conditions — Esophagitis, Peptic | interventions — Rabeprazole; Lansoprazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Rabeprazole (Experimental): Rabeprazole 20 mg tablet orally once daily before breakfast for 28 to 56 days.
  Interventions: Drug: Rabeprazole
- Lansoprazole (Active Comparator): Lansoprazole 30 mg capsule orally once daily before breakfast for 28 to 56 days.
  Interventions: Drug: Lansoprazole

INTERVENTIONS:
Drug: Rabeprazole — Rabeprazole 20 mg tablet orally once daily before breakfast for 28 to 56 days.
  Arms: Rabeprazole
Drug: Lansoprazole — Lansoprazole 30 mg capsule orally once daily before breakfast for 28 to 56 days.
  Arms: Lansoprazole

SUMMARY:
The purpose of this study is to compare the treatment effects of rabeprazole and lansoprazole depending on the genotyping (process of determining the genetic constitution) of CYP2C19 in treating reflux esophagitis (caused by gastroesophageal reflux; deterioration of the protective lining on the inner wall of the lower esophagus); and to evaluate the cure rate of reflux esophagitis on endoscopy (a thin flexible tube with a microscopic camera at the end which is passed down your throat into the esophagus, stomach, and duodenum) after treatment with rabeprazole and lansoprazole.

DETAILED DESCRIPTION:
This is a prospective (study following participants forward in time), open-label (all people know the identity of the intervention), multi-center (conducted in more than 1 center), randomized (study drug assigned by chance) study in participants with reflux esophagitis. The study will include 4 visits: Visit 1 (Screening period of up to 14 days), Visit 2 (Day 1), Visit 3 (Day 29+3), and Visit 4 (Day 56). After Screening, eligible participants will be analyzed on Visit 2 (Day 1) for symptoms during past week, At visit 3 (Day 29+3) participants will be randomly assigned to 1 of the 2 treatment groups: rabeprazole 20 milligram (mg) or lansoprazole 30 mg group. Participants will receive rabeprazole 20 mg tablet orally once daily for 28 to 56 days or lansoprazole 30 mg capsule orally once daily for 28 to 56 days. A post-study follow-up visit will be conducted only if participant will be affected by any serious adverse event within 30 days after the completion of study drug. Participants will primarily be assessed for the cure rate of reflux esophagitis based on endoscopy of 2 groups. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with reflux esophagitis of Grade A or higher by Los Angeles (LA) classification based on the endoscopy among participants complaining of gastroesophageal reflux symptoms (such as: Heartburn, regurgitation, globus sensation, chronic [lasting a long time] cough [sudden, loud flow if air from the lungs], epigastric [area above the navel] pain, non-cardiac chest pain, hoarseness, or dysphagia), or those who diagnosed with reflux esophagitis of Grade B or higher without complaining of symptoms
* Participants without other serious disease except the study indication (reflux esophagitis)
* Participants with hematology (related to blood) panel, serum chemistry panel, or urinalysis result clinically within twice the normal range
* Female Participants of child-bearing potential who are using the appropriate contraceptive or with a negative urine pregnancy test

Exclusion Criteria:

* Participants with other serious gastrointestinal disease except reflux esophagitis (example: digestive tract cancer [abnormal tissue that grows and spreads in the body until it kills], hepatic disease, pancreatic disease, and ulcer. However, the scar of an ulcer is included in study targets
* Participants with other serious concomitant disease(s) such as renal disorder, cerebrovascular disease, cardiovascular disease, hepatic disease, and severe respiratory disease
* Participants with medical history of upper gastrointestinal tract surgery, esophagostenosis, or a chalasia
* Participants with hematology panel, serum chemistry panel, or urinalysis result of above twice the normal range
* Participants who cannot discontinue proton pump inhibitors or Histamine 2 antagonist which may have influence on the study, 4 weeks before the start of this clinical study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2007-05; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Korea, Ltd., Korea Clinical Trial, Study Director — Janssen Korea, Ltd., Korea

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Out of 225 participants consented, 217 were assigned to the study medication.
Groups:
- Rabeprazole: Rabeprazole 20 milligram (mg) tablet orally once daily before breakfast for 28 to 56 days
Period: Overall Study
Arm/Group | Rabeprazole | Lansoprazole
Started | 108 | 109
Completed | 91 | 92
Not Completed | 17 | 17
Not completed — Participant's evasion of hospital visit | 5 | 4
Not completed — Withdrawal by Subject | 2 | 4
Not completed — Physician Decision | 5 | 1
Not completed — Adverse Event | 1 | 0
Not completed — Participants' non-cooperation | 2 | 3
Not completed — Other | 2 | 3
Not completed — Other | 0 | 2

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were measured for full analysis set (FAS) population. It included participants who received study medication at least once and had follow-up data that could be used after Baseline among participants who met eligibility criteria. Last observation carried forward (LOCF) was used.
Groups:
- Total: Total of all reporting groups
Arm/Group | Rabeprazole | Lansoprazole | Total
Number analyzed (Participants) | 87 | 91 | 178
Age Continuous [Mean (Standard Deviation); unit: Years] — Age continuous was measured for full analysis set (FAS) population. It included participants who received study medication at least once and had follow-up data that could be used after Baseline among participants who met eligibilitycriteria. Last observation carried forward (LOCF) was used.
  Years | 49.70 (11.72) | 49.74 (12.65) | 49.72 (12.17)
Sex: Female, Male [Count of Participants; unit: Participants] — Gender is measured for the FAS popluation. It included participants who received study medication at least once and had follow-up data that could be used after Baseline among participants who met eligibilitycriteria. Last observation carried forward (LOCF) was used.
  Participants
    Female | 12 | 22 | 34
    Male | 75 | 69 | 144

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Completely Cured of Reflux Esophagitis Evaluated by Endoscopy Based on CYP2C19
Description: Reflux esophagitis evaluated by endoscopy as per LA Classification graded as: A=1 or more mucosal breaks no longer than 5 millimeter (mm) that did not extend between tops of 2 mucosal folds, B=1 or more mucosal breaks more than 5 mm long that did not extend between tops of 2 mucosal folds, C=1 or more mucosal break continuous between the tops of 2 or more mucosal folds but involves less than 75 percent of circumference, D=1 or more mucosal break involving at least 75 percent of circumference. Participants that were not categorized in any of the above mentioned grades (A to D) were considered as cured of reflux esophagitis. Participants were classified as CYP2C19 homozygous extensive, heterozygous extensive and poor metabolizers.
Time Frame: Day 57
Population: The Full analysis set (FAS) included participants who received study medication at least once and had follow-up data that could be used after Baseline among participants who met eligibility criteria. Last observation carried forward (LOCF) was used. Here, 'n'=participants evaluated for particular category of this outcome measure.
Measure: Number; unit: Percentage of participants
Arm/Group | Rabeprazole | Lansoprazole
Number analyzed (Participants) | 87 | 91
Percentage of participants
  Homozygous Extensive Metabolizer (n=42, 35) | 97.37 | 93.94
  Heterozygous Extensive Metabolizer (n=30, 38) | 100.00 | 100.00
  Poor Metabolizer (n=15, 18) | 93.33 | 100.00
Statistical Analysis 1: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.8849, Chi-squared — Homozygous extensive metabolizer
Statistical Analysis 2: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.8650, Chi-squared — Heterozygous extensive metabolizer
Statistical Analysis 3: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.2660, Chi-squared — Poor metabolizer

2. Secondary Outcome: Change From Baseline in Symptoms of Reflux Esophagitis Evaluated by the Symptom Assessment Questionnaire
Description: Gastroesophageal reflux disease and abdominal GI-related symptoms (heartburn, regurgitation, globus sensation, chronic cough, epigastric pain, non cardiac chest pain, hoarseness, dysphagia, abdominal distension, bloating, post-prandial discomfort, early satiety, nausea, vomiting, belching) experienced by participants were assessed and graded into 4 categories: 0 (Nothing)=No symptom, 1 (Mild)=A little but not uncomfortable, 2 (Moderate)=Present but interfering daily life activities a little, 3 (Severe)=Very uncomfortable, interfering daily life activities or sleeping.
Time Frame: Baseline and Day 57
Population: The FAS included participants who received study medication at least once and had follow-up data that could be used after Baseline among participants who met eligibility criteria. Last observation carried forward (LOCF) was used. Here, 'n'=participants evaluated for particular category of this outcome measure
Measure: Mean (Standard Deviation); unit: Units on a scale
Groups:
- Lansoprazole: Lansoprazole group 30 mg capsule orally once daily before breakfast for 28 to 56 days
Arm/Group | Rabeprazole | Lansoprazole
Number analyzed (Participants) | 87 | 91
Units on a scale
  Baseline: Heartburn (n=87, 91) | 0.61 (0.84) | 0.59 (0.89)
  Baseline:Regurgitation (n=87, 91) | 0.98 (0.93) | 0.93 (0.96)
  Baseline: Globus sensation (n=87, 91) | 0.55 (0.82) | 0.82 (0.78)
  Baseline: Chronic cough (n=87, 91) | 0.34 (0.70) | 0.30 (0.66)
  Baseline: Epigastric pain (n=87, 90) | 0.91 (1.00) | 0.94 (0.95)
  Baseline: Non cardiac chest pain (n=85, 90) | 0.33 (0.71) | 0.26 (0.66)
  Baseline: Hoarseness (n=87, 90) | 0.23 (0.54) | 0.22 (0.54)
  Baseline: Dysphagia (n=87, 91) | 0.16 (0.50) | 0.22 (0.57)
  Baseline: Abdominal distension (n=87, 91) | 0.61 (0.84) | 0.59 (0.80)
  Baseline: Bloating (n=87, 90) | 0.55 (0.82) | 0.44 (0.75)
  Baseline: Post-prandial discomfort (n=87, 91) | 0.53 (0.78) | 0.55 (0.76)
  Baseline: Early satiety (n=86, 91) | 0.27 (0.58) | 0.25 (0.55)
  Baseline: Nausea (n=87, 91) | 0.16 (0.48) | 0.13 (0.37)
  Baseline: Vomiting (n=87, 91) | 0.08 (0.38) | 0.02 (0.15)
  Baseline: Belching (n=87, 91) | 0.38 (0.70) | 0.36 (0.62)
  Change at Day 57: Heartburn (n=87, 91) | -0.55 (0.83) | -0.54 (0.90)
  Change at Day 57: Regurgitation (n=87, 91) | -0.89 (0.93) | -0.84 (0.95)
  Change at Day 57: Globus sensation (n=87, 91) | -0.31 (0.69) | -0.32 (0.66)
  Change at Day 57: Chronic cough (n=87, 91) | -0.22 (0.64) | -0.21 (0.61)
  Change at Day 57: Epigastric pain (n=87, 90) | -0.77 (0.95) | -0.77 (0.92)
  Change at Day 57:Non cardiac chest pain (n=85, 90) | -0.28 (0.65) | -0.20 (0.54)
  Change at Day 57: Hoarseness (n=87, 90) | -0.14 (0.51) | -0.17 (0.55)
  Change at Day 57: Dysphagia (n=87, 91) | -0.11 (0.44) | -0.14 (0.48)
  Change at Day 57: Abdominal distension (n=87, 91) | -0.38 (0.80) | -0.40 (0.76)
  Change at Day 57: Bloating (n=87, 90) | -0.41 (0.72) | -0.37 (0.69)
  Change at Day57:Post-prandial discomfort (n=87,91) | -0.45 (0.73) | -0.35 (0.74)
  Change at Day 57: Early satiety (n=86, 91) | -0.21 (0.49) | -0.16 (0.58)
  Change at Day 57: Nausea (n=87, 91) | -0.16 (0.48) | -0.11 (0.38)
  Change at Day 57: Vomiting (n=87, 91) | -0.08 (0.38) | -0.02 (0.15)
  Change at Day 57: Belching (n=87, 91) | -0.25 (0.70) | -0.29 (0.54)
Statistical Analysis 1: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.7734, Wilcoxon rank-sum test — Change at Day 57: Heartburn
Statistical Analysis 2: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.6414, Wilcoxon rank-sum test — Change at Day 57: Regurgitation
Statistical Analysis 3: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.7809, Wilcoxon rank-sum test — Change at Day 57: Globus sensation
Statistical Analysis 4: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.8294, Wilcoxon rank-sum test — Change at Day 57: Chronic cough
Statistical Analysis 5: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.9874, Wilcoxon rank-sum test — Change at Day 57: Epigastric pain
Statistical Analysis 6: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.2776, Wilcoxon rank-sum test — Change at Day 57: Non cardiac chest pain
Statistical Analysis 7: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.6295, Wilcoxon rank-sum test — Change at Day 57: Hoarseness
Statistical Analysis 8: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.5335, Wilcoxon rank-sum test — Change at Day 57: Dysphagia
Statistical Analysis 9: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.8068, Wilcoxon rank-sum test — Change at Day 57: Abdominal distension
Statistical Analysis 10: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.5680, Wilcoxon rank-sum test — Change at Day 57: Bloating
Statistical Analysis 11: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.5913, Wilcoxon rank-sum test — Change at Day 57: Post-prandial discomfort
Statistical Analysis 12: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.5566, Wilcoxon rank-sum test — Change at Day 57: Early satiety
Statistical Analysis 13: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.7047, Wilcoxon rank-sum test — Change at Day 57: Nausea
Statistical Analysis 14: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.3654, Wilcoxon rank-sum test — Change at Day 57: Vomitting
Statistical Analysis 15: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.5310, Wilcoxon rank-sum test — Change at Day 57: Belching

3. Secondary Outcome: Overall Assessment of Study Medication by Investigator
Description: Investigator's overall assessment of study medication based on the global symptom assessment was measured. The assessment was categorized as: 2=very good, 1=good, 0=as usual, -1=bad and -2=very bad.
Time Frame: Day 57
Population: The FAS included participants who received the study medication at least once and had follow-up data that could be used after the Baseline among the participants meeting the eligibility criteria of this study. LOCF was used. Here, 'N'=participants evaluated for this outcome measure.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Rabeprazole | Lansoprazole
Number analyzed (Participants) | 84 | 89
Units on a scale | 1.37 (0.71) | 1.43 (0.74)
Statistical Analysis 1: Comparison: Rabeprazole vs Lansoprazole; Test type: Superiority or Other; p = 0.5032, Wilcoxon rank-sum test

ADVERSE EVENTS:
Time Frame: Baseline up to Day 57
Arm/Group | Rabeprazole | Lansoprazole
Serious Adverse Events (participants affected / at risk) | 2/108 | 0/109
Other Adverse Events (participants affected / at risk) | 42/108 | 42/109
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole (N=108) | Lansoprazole (N=109)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0
Haemorrhoid operation (Surgical and medical procedures) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rabeprazole (N=108) | Lansoprazole (N=109)
Abdominal distension (Gastrointestinal disorders) | 19 | 18
Abdominal pain (Gastrointestinal disorders) | 12 | 17
Dyspepsia (Gastrointestinal disorders) | 10 | 15
Abdominal pain upper (Gastrointestinal disorders) | 9 | 12
Dysphagia (Gastrointestinal disorders) | 10 | 10
Nausea (Gastrointestinal disorders) | 8 | 9
Regurgitation (Gastrointestinal disorders) | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 4 | 0
Sensation of foreign body (General disorders) | 13 | 16
Early satiety (General disorders) | 11 | 11
Non-cardiac chest pain (General disorders) | 6 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 18 | 15
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 9 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No